CLINICAL TRIAL: NCT01182519
Title: Association of Smoking, Lung Inflammation and Lung Metastases From Breast Cancer
Brief Title: Lung Inflammation and Lung Metastases From Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Other Study IDs: 10-115
Record Dates: First submitted 2010-08-13; First posted 2010-08-16 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: lung inflammation; lung metastases; 10-115
MeSH Terms: conditions — Breast Neoplasms; Pneumonia | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and Blood

GROUPS / COHORTS (2):
- Diagnosed with metastatic breast cancer: The primary objective of this study is to examine the association between urinary PGE-M and the presence or absence of lung metastases in patients with breast cancer. These patients will be subdivided into a set with lung metastases (group 1A; clinically assessed as per guidelines below) versus those with no evidence of lung metastases (group 1B; "no known lung metastases"). Group #2 (control) will have been treated for early stage breast cancer and will have no known metastases.
  Interventions: Behavioral: questionnaire, blood draw and urine sample
- History of early breast cancer: History of early breast cancer and currently no evidence of disease
  Interventions: Behavioral: questionnaire, blood draw and urine sample

INTERVENTIONS:
Behavioral: questionnaire, blood draw and urine sample — Patients will be asked to participate on a single day. After study registration they will be asked to complete the questionnaire. All participants will complete a questionnaire detailing tobacco and NSAID exposure, as well as detailing any other inflammatory conditions of the lung. Then the patient will give a single blood sample (up to 3 tubes) and a single urine sample.

SUMMARY:
The purpose of this study is to find out if there is a link between cigarette smoking, inflammation and the spread of breast cancer to the lung. We think that women who are current or former smokers may be at increased risk for breast cancer spreading to the lung compared to women who have never smoked. Smoking causes inflammation in the lung in some women. Researchers at Memorial Sloan-Kettering (MSKCC) think that smoking-related lung inflammation may increase the chance of breast cancer spreading to the lung. In order to find out whether inflammation plays a role in breast cancer spreading to the lung, we will measure a urinary marker of lung inflammation. This will allow us to determine if this marker is more commonly elevated in women with breast cancer that has spread to the lung compared to those without breast cancer in the lung. We will also collect DNA from blood to have the opportunity to determine if there are differences in DNA in women with or without breast cancer that has spread to the other sites including the lung. We will also collect blood to determine if we can identify risk factors for the spread of breast cancer to the lungs.

ELIGIBILITY:
Inclusion Criteria:

* Registered patient at MSKCC
* Histologically proven breast cancer. It is not necessary that pathology be reviewed at MSKCC
* Age ≥18 years Group 1 (A and B)
* Diagnosed with metastatic breast cancer on biopsy or imaging study.
* Patients will be considered to have lung metastases, and will be assigned to group 1A if any of the following criteria are met, otherwise patients will be assigned to group 1B "No known Lung Metastases," Biopsy-proven lung metastasis.
* Pleural effusion with cytologic evidence of malignancy.
* Pleural effusion, exudative in character, without alternative explanation and attributed, in the opinion of the clinician to metastatic disease.
* Symptoms attributable to lung metastases and a radiological pattern interpreted by a radiologist as suspicious for metastatic disease.
* Any pulmonary nodule on chest radiograph, CT scan, PET-CT or MRI, which is interpreted by the clinician and radiologist to be metastatic in etiology, whether or not a biopsy was performed, and regardless of symptoms.
* A radiographic pattern interpreted by a radiologist as consistent with lymphangitic carcinomatosis.

Group 2 (Controls)

* History of early breast cancer and currently no evidence of disease

Exclusion Criteria:

* Inability to provide written informed consent.
* Inability to complete smoking and NSAID questionnaire.
* Steroid use within the previous 4 weeks.
* Radiotherapy to the breast, chest wall or axilla within the previous 3 months.
* Men with breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the above inclusion and exclusion criteria will be approached by a member of the study team and be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The association between urinary PGE-M and the presence or absence of lung metastases | 2 years
  in patients with breast cancer

SECONDARY OUTCOMES:
The putative link between smoking and site-specific metastases from breast cancer | 2 years
Polymorphisms for genes linked to inflammation (germ line DNA SNPs) | 2 years
  with the presence or absence of lung metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Hudis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm